CLINICAL TRIAL: NCT03808948
Title: Estimating Versus Measuring Plasma Volume and Kidney Function in Acute Decompensated Congestive Heart Failure (EMPaKT-CHF)
Brief Title: FAST PV and mGFR™ Technology in Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: FAST BioMedical (Industry)
Responsible Party: Principal Investigator, Kai Schmidt-Ott, Principal Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EmPaKt-CHF; 2018-002638-18 (EudraCT Number)
Record Dates: First submitted 2019-01-08; First posted 2019-01-18 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: CHF
Keywords: congestive heart failure; glomerular filtration rate; plasma volume
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All Patients (Experimental): VFI dose: 47 mg / 3 mL Number of doses: 2 Route of administration: intravenous
  Interventions: Device: VFI

INTERVENTIONS:
Device: VFI — The IV-administered visible fluorescent injectate (VFI)™ agent comprises a mixture of 2 different molecular weight carboxymethyl dextran molecules (5 kD and 150 kD) with different fluorescent dye molecules attached.

SUMMARY:
This is an investigator-initiated, one-armed, phase 2 clinical trial using an injectable fluorescent tracer to assay and evaluate measured plasma volume (mPV) and measured glomerular filtration rate (mGFR) in hospitalized patients with acute decompensated congestive heart failure (CHF).

DETAILED DESCRIPTION:
This investigator-initiated, one-armed study is designed to evaluate the safety and function of the FAST PV and mGFR Technology in patients with CHF. Data from the FAST PV and mGFR Technology will not be evaluable by the treating physician, but will be made available to the study investigators and to an adjudication committee.

Patients enrolled in the study will be administered the VFI (Day 1) and with a second dose occurring 24-48 hours after the initial dose (Day 3).

After consenting to be enrolled in the study, patients meeting the enrollment criteria will receive a single dose of two component VFI. Blood draws (3 mL) will be collected pre-dose and at 15, 30, 60, and 180 minutes post-dose, which will be subsequently used to determine the patient's blood volume and mGFR using the FAST PV and mGFR Technology. Patients will be treated according to standard of care throughout the time of their hospitalization. A second dose of VFI will be administered 48 (+/- 5) hours after the initial dosing. Again, blood draws (3 mL) will be collected pre-dose and at 15, 30, 60, and 180 minutes post-dose. Plasma volume (PV) was determined using the average concentrations of the higher molecular marker of VFI of the early 15 min and the 60 min time point. The concentration of the small dextran GFR marker at time zero was back calculated from the measured PV by dividing the known dose into the measured PV. The time points were then fitted using atwo-compartment model and the resulting area under the curve was calculated. The use of the time point 0 determination helped to better resolve the shape of the clearance curve.

Study-related blood samples will be obtained on days 1, 2, 3, 4, and 5 to measure serum creatinine (days 1-5), hematocrit (days 1, 3), and N-terminal pro-brain natriuretic peptide (NT-pro-BNP), creatine phosphokinase (CPK), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, bilirubin total and direct, and international normalized ratio (INR) (days 1, 3, and 5); and will be stored for future testing of additional parameters in the research fields of acute decompensated heart failure and acute kidney injury.

The available laboratory values will be entered in the Dosing Day Case Report Form (CRF), along with any copies of physician's notes and orders entered that day. Prior to administering the first and second dose of VFI, the physician will be asked to complete a very brief survey to provide a qualitative assessment of the patient's perceived volume status and renal function prior to initiating the FAST PV and mGFR measurements.

Laboratory values and assessments will be captured on each day that the VFI is administered, and these data will be entered into the CRF. Any adverse events (AEs) determined by the investigator to be related or possibly related to the VFI will be captured. Patients will receive a followup phone call 7 days (± 2 days) after the first dose of VFI was administered, and a second follow up call 30 days after the first dose of VFI was administered as an end of study (EOS) follow up call. Any AEs determined by the investigator will be captured during the follow up calls and will be followed to resolution. Additionally, in-person follow-up visits may be scheduled as needed.

Upon conclusion of the study, the recorded clinical data will be provided to an independent data adjudication committee (DAC) in a pseudonymized fashion. The DAC will be asked to review the available data at the time of the first dosing, and the measured GFR and PV data for the first dosing day will be provided. The DAC will then be asked to fill out a survey asking whether the mGFR and PV data would have influenced their treatment decision, and if so, indicate what they would have done differently.

Following the evaluation of mGFR and PV data at the time of the initial VFI dose, the mGFR and PV data determined from the second VFI dosing point will be provided to the DAC. The DAC will then be asked to fill out a separate survey asking how the actual measured PV and GFR differ from the clinical assessments, whether the mGFR and PV data would influence their treatment decision, and if so, indicate what they would have done differently.

After all assessments have been completed, the DAC will review the results of their analyses and compile a summary report on the secondary endpoints as well as their assessment of the overall impact of the PV and mGFR on clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent indicating an understanding of the purpose of and procedures required for the study and willingness to participate in the study prior to any study-related measures present.
* Hospitalized patient with acute decompensated heart failure, diagnosed on the basis of the presence of at least one symptom (dyspnea, orthopnea, or edema) and one sign (rales, peripheral edema, ascites, or pulmonary vascular congestion on chest radiography) of heart failure.
* ≥ 18 years of age.
* Male with female partners of childbearing potential give agreement to practice abstinence or use condoms from enrollment through 90 days after administration of the last dose of study drug present.
* Partner of a male patient: Agreement to use a medically acceptable method of contraception (a barrier method, intrauterine device, or hormonal contraception) from enrollment through 90 days after administration of the last dose of study drug present.
* Male patient agrees to not donate sperm from enrollment through 90 days after administration of the last dose of study drug present.
* A female patient is eligible to enter the study if she is not pregnant or nursing; of non-childbearing potential (ie, post-menopausal defined as having been amenorrheic for at least 1 year prior to screening, or has had bilateral tubal ligation at least 6 months prior to administration of study drug or bilateral oophorectomy or complete hysterectomy); and if of childbearing potential, must have a negative urine or serum pregnancy test within 24 h prior to drug administration and be using a highly effective means of contraception during study participation and until 1 month after the last dose of study drug. Highly effective contraception methods include total abstinence or combination of any two of the following: (i) use of oral, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy; (ii) placement of an intrauterine device (IUD) or intrauterine system (IUS); and (iii) barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps). In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
* Patient is able to communicate effectively with the study personnel.
* Patient is informed of the nature and risks of the study and give written informed consent prior to enrollment.

Exclusion Criteria:

* New or ongoing myocardial infarction or unstable angina present at the time of planned study inclusion.
* Patient shows evidence of severe infection other than pneumonia, or active internal bleeding (characterized by recent decrease of blood hemoglobin concentration by more than 2 g/dl).
* Patient experiences new onset atrial fibrillation.
* Patient has an elective surgery planned during the 30 days he/she is enrolled in the study.
* Patient has a psychiatric disease or a history of illicit drug use that would prohibit him/her from complying with study requirements.
* Prior exposure to VFI present.
* History of any clinically significant allergic or negative reactions, side effects, or anaphylaxis to fluorescent dyes, or dextran molecules present.
* Patient requires intravenous vasodilators or inotropic agents (other than digoxin or digitoxin) for heart failure.
* Patient undergoes chronic dialysis (for example peritoneal or hemodialysis) treatments.
* Patient is in cardiogenic shock or on vasopressors.
* Hypotension as defined by blood pressure ≤ 90 mm Hg systolic and/or ≤ 50 mm Hg diastolic exists.
* Patient has significant non-cardiac disease of other organ system (eg, malignancies, significant neurological disease).
* Patient does not have a working telephone.
* Patient is pregnant or nursing (lactating), where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Lack of willingness to storage and disclosure of pseudonymous disease data in the context of the clinical trial present.
* Patient has a participation in another interventional clinical trial during this study or within 30 days (or longer) before entry into this study (as a minimum; 5 x elimination half-life / terminal elimination of an investigational medicinal product).
* Patient is legally detained in an official institution.
* Patient is dependent on the sponsor, the investigator, or the trial sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-08-17 (Actual); Study Completion 2019-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai M Schmidt-Ott, Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hinze C, Karaiskos N, Boltengagen A, Walentin K, Redo K, Himmerkus N, Bleich M, Potter SS, Potter AS, Eckardt KU, Kocks C, Rajewsky N, Schmidt-Ott KM. Kidney Single-cell Transcriptomes Predict Spatial Corticomedullary Gene Expression and Tissue Osmolality Gradients. J Am Soc Nephrol. 2021 Feb;32(2):291-306. doi: 10.1681/ASN.2020070930. Epub 2020 Nov 25. PMID 33239393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A totally of 50 hospitalized patients were enrolled between January 10th, 2019 and August 15th, 2019.
Pre-assignment Details: No patients were excluded after enrollment but before assignment to the treatment group.
Period: Overall Study
Arm/Group | All Patients
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 50
Weight day 1 (kg) [Mean (Standard Deviation); unit: kilograms] | 89.21 (22.24)
Height day 1 (cm) [Mean (Standard Deviation); unit: Centimeters] | 172.84 (10.62)
BMI day 1 (kg/m2) [Mean (Standard Deviation); unit: Kilograms / meter squared] | 29.7 (6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related AEs and Serious Adverse Events (SAEs)
Description: The percentage of treatment emergent SAEs considered to be surely related to the VFI should be zero.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 50
Participants | 0

2. Primary Outcome: Percentage Difference in Mean Plasma Concentration of FD003 Over the 15-, 30-, and 60-minute Blood Draws on Days 1 and 3
Description: Function of the FAST PV measurement will be assessed by determining the plasma stability of the FD003 high molecular weight marker over the 15, 30, and 60 minute blood draws and applying the following criteria:
  * The FAST PV measurement is considered as stable, if the mean plasma concentration of FD003 at 30 minutes is not more than 10% lower than the mean plasma concentration at 15 minutes AND if the mean plasma concentration at 60 minutes is not more than 10% lower than the mean plasma concentration at 30 minutes
  * We will determine the percentage of patients which show a decline in the plasma concentration of FD003 of more than 10% from 15min to 30min and separately from 30 min to 60min. This percentage should be ideally close to 0.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Percent difference, plasma concentration
Arm/Group | All Patients
Number analyzed (Participants) | 50
Percent difference, plasma concentration
  Difference between Day 1 mean plasma concentration of FD003 at 15 minutes and 30 minutes | -2.36 (7.94)
  Difference between Day 3 mean plasma concentration of FD003 at 15 minutes and 30 minutes | -3.12 (11.29)
  % difference between Day 1 mean plasma concentration of FD003 at 30 minutes and 60 minutes | -0.8 (5.6)
  % difference between Day 3 mean plasma concentration of FD003 at 30 minutes and 60 minutes | -0.79 (8.67)

3. Secondary Outcome: Accuracy Between Estimated PV (ePV) on Days 1 and 3 (by Established Measures) and Measured PV (mPV; as Assessed by FAST Methodology) Defined as the Percentage of the Population With a <15% and <30% Difference Between ePV and mPV
Description: The percentage difference between ePV and mPV were evaluated to consider the percentage of the population with a <15% and <30% difference between ePV and mPV on day 1 and day 3
Time Frame: 3 days
Population: One patient did not have a hematocrit available for ePV determination, fourteen patients did not have day 3 measurements of mPV.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 49
Participants
  Number patients where ePV (Kaplan Hakim) was within 15% of mPV day1 | 32
  Number patients where ePV (Kaplan Hakim) was within 30% of mPV day 1 | 44
  Number patients where ePV (Kaplan Hakim) was within 15% of mPV day3: number analyzed (Participants) | 36
  Number patients where ePV (Kaplan Hakim) was within 15% of mPV day3 | 24
  Number patients where ePV (Kaplan Hakim) was within 30% of mPV day3: number analyzed (Participants) | 36
  Number patients where ePV (Kaplan Hakim) was within 30% of mPV day3 | 30

4. Secondary Outcome: Accuracy Between Estimated Total Blood Volume (TBV) on Days 1 and 3 and Measured TBV (mTBV; Calculated From mPV and Measured Hematocrit) Defined as the Percentage of the Population With a <15% and <30% Difference Between ePV and mPV
Description: Accuracy between the Nadler's Formula as an estimate of total blood volume (TBV) and measured blood volume (mTBV) on days 1 and 3 as determined by the percentage of the population with a <15% and <30% difference between ePV and mPV
Time Frame: 3 days
Population: One patient did not have a hematocrit on day 1 for calculation of mTBV and eTBV, twelve patients did not receive a second measurement on day 3, two patients that recieved a second measurement, did not have a hematocrit on day 3 for calculation of mTBV and eTBV
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 49
Participants
  Number of patients where eTBV was within 15% of mTBV value day1 | 32
  Number of patients where eTBV was within 30% of mTBV value day1 | 45
  Number of patients where eTBV was within 15% of mTBV value day3: number analyzed (Participants) | 36
  Number of patients where eTBV was within 15% of mTBV value day3 | 25
  Number of patients where eTBV was within 30% of mTBV value day3: number analyzed (Participants) | 36
  Number of patients where eTBV was within 30% of mTBV value day3 | 32

5. Secondary Outcome: Accuracy of eGFR Determined by CKD-EPI-SCr and mGFR on Day 1 and Day 3 Defined the Percentage of the Population With a <15% and <30% Difference Between eGFR and mGFR
Description: To evaluate whether estimated Glomerular Filtration Rate (eGFR) (calculation by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula) on days 1 and 3 provides an accurate estimate of measured GFR (mGFR; assessed by FAST methodology) in heart failure patients under-going active fluid management, determined by the percentage of patients with a <15% and <30% difference between eGFR and mGFR
Time Frame: 3 days
Population: twelve patients did not have mGFR measurement on day 3, so only 38 patients are analyzed on day 3
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 50
Participants
  Number of patients where eGFR was within 15% of mGFR value on Day 1. | 20
  Number of patients where eGFR was within 15% of mGFR value on Day 3.: number analyzed (Participants) | 38
  Number of patients where eGFR was within 15% of mGFR value on Day 3. | 10
  Number of patients where eGFR was within 30% of mGFR value on Day 1. | 33
  Number of patients where eGFR was within 30% of mGFR value on Day 3.: number analyzed (Participants) | 38
  Number of patients where eGFR was within 30% of mGFR value on Day 3. | 24

6. Secondary Outcome: Percentage of the Population That Developed Acute Kidney Injury (AKI) Within the Following 48-72 Hour and Prediction of AKI by mGFR/eGFR Ratio on Days 1 and 3
Description: To evaluate the percentage of patients developing acute kidney injury (AKI) within the following 48-72 hours on day 1 and day 3 and to evaluate whether patients with a low mGFR/eGFR ratio on days 1 and 3 are at higher risk of developing acute kidney injury (AKI) within the following 48-72 hours using a binary logisitic regression with AKI as binary outcome and mGFR/eGFR as independent variate
Time Frame: 48-72h
Population: 36 patients had data for AKI determination 48h after day 1, 32 patients had data for AKI determination after day 3
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 36
Participants
  Number of patients with AKI within 48h after day 1 | 17
  Number of patients with AKI within 48h after day 3: number analyzed (Participants) | 32
  Number of patients with AKI within 48h after day 3 | 11
Statistical Analysis 1: Comparison: All Patients; Binary logistic regression with mGFR/eGFR ratio as independent variate, AKI as binary outcome; Test type: Other; p = 0.4842, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.08 to 1.97]

7. Secondary Outcome: Percentage of Patients Who Are Refractory to Diuretic Therapy
Description: Being refractory to diuretic therapy (defined as any dosage increases of furosemide i.v. dose equivalent, adding thiazide after day 1, requirement of ultrafiltration/RRT within the next 24-48 hours, failure to improve subjectively in PGA and dyspnoea scales, failure of mean weight loss during the study period Day 1-Day 5 of at least 0,5 kg/d).
Time Frame: 5 days
Population: one patient did not have weight data, two patients were discharged after first measurement (day 1) so no lineary observation was possible
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 47
Participants
  Not refractory to diuretics | 7
  Refractory to diuretics | 40

8. Secondary Outcome: Percentage of Population in Which Clinical Decision Making Would Have Been Influenced by Adding FAST GFR and PV Measurements to Clinical Routine Determined by Survey Response (by an Adjudication Committee)
Description: Percentage of patients for whom the data decision committee decided to increase or decrease the dose of diuretics, guideline-directed medical therapy (GDMT), beta-blockers, or RAAS inhibitors from the dose indicated by the treating physician after considering the mPV/mTBV determined using FAST BioMedical technology.
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 50
Participants
  Number or patients where adjudication committee would have changed diuretic dose | 40
  Number or patients where adjudication committee would have changed RAASi dose | 5
  Number or patients where adjudication committee would have changed beta blocker dose | 6
  Number or patients where adjudication committee would have changed GDMT | 1

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 21/50
Other Adverse Events (participants affected / at risk) | 37/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=50)
Pneumonia (Infections and infestations) | 3
Endocarditis (Infections and infestations) | 2
Infectious pleural effusion (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative delirium (Injury, poisoning and procedural complications) | 1
cardiac failure (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Acute kidney Injury (Renal and urinary disorders) | 3
Azotaemia (Renal and urinary disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Ischaemia (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Troponin increased (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=50)
Diarrhoea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1
Varices oesophageal (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Pneumonia (Infections and infestations) | 6
Endocarditis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis rotavirus (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Troponin increased (Investigations) | 2
Bilirubin conjugated increased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatine phosphokinase abnormal (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Brain natriuretic peptide increased (Investigations) | 1
Procalcitonin abnormal (Investigations) | 1
Procalcitonin increased (Investigations) | 1
Pyrexia (General disorders) | 3
Chest pain (General disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pain (General disorders) | 1
Xerosis (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 3
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative delirium (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Cardiac failure (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Sleep disorder (Psychiatric disorders) | 5
Delirium (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Azotaemia (Renal and urinary disorders) | 1
End stage renal disease (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Ischaemia (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Penile haemorrhage (Reproductive system and breast disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Phimosis (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Immobile (Social circumstances) | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT03808948/Prot_002.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT03808948/SAP_001.pdf